CLINICAL TRIAL: NCT05884970
Title: In Vivo Efficacy of Salbutamol (Sandoz) Versus Salbutamol Ventolin (GSK) in Children With Asthma
Acronym: Salsa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Principal Investigator, Ellen Croonen, dr. E Croonen, Principal Investigator, Canisius-Wilhelmina Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL67238.091.19
Record Dates: First submitted 2023-03-30; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Agents, Anti Asthmatic; Asthma in Children
Keywords: albuterol; ventolin; salbutamol; sandoz

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- FEV1 >90% (Active Comparator): Children with lung function FEV1 > 90%
  Interventions: Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK"
- FEV1 80-90% (Active Comparator): Children with lung function FEV1 80-90%
  Interventions: Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK"
- FEV1 70-80% (Active Comparator): Children with lung function FEV1 70-80%
  Interventions: Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK"
- FEV1 60-70% (Active Comparator): Children with lung function FEV1 60-70%
  Interventions: Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK"
- FEV1 < 60% (Active Comparator): Children with lung function FEV1 < 60%
  Interventions: Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz"; Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK"

INTERVENTIONS:
Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Sandoz" — Efficacy of Salbutamol Sandoz will be compared to Salbutamol Ventolin GSK (reference)
Drug: "100 mcg Salbutamol Sandoz" and "300 mcg Salbutamol Ventolin GSK" — Efficacy of Salbutamol Sandoz will be compared to Salbutamol Ventolin GSK (reference)
Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Sandoz" — Efficacy of Salbutamol Sandoz will be compared to Salbutamol Ventolin GSK (reference)
Drug: "100 mcg Salbutamol Ventolin GSK" and "300 mcg Salbutamol Ventolin GSK" — Efficacy of Salbutamol Sandoz will be compared to Salbutamol Ventolin GSK (reference)

SUMMARY:
In this study, the investigators hypothesize that the reference product (SalbR/Ventolin) is more effective than SalbG (Salbutamol Sandoz) at improving the lung function in children with asthma, and that this difference increases alongside the severity of the airway resistance. (Null hypothesis: There is no difference).

This could be explained by different properties and deposition of the aerosol.

Purpose of this research:

Rejecting the null hypothesis. This is based on the answers to the questions below.

Research questions:

1. Is there a difference between the increase in FEV1 (and FVC) after 100 μg SalbG versus FEV1 after 100 μg SalbR in children aged 4-14 years with insufficient asthma control? (primary question)
2. Is there a difference in the subjective feeling of the children after inhalation with 100 μg SalbR and after 100 μg SalbG, measured with a VAS score?
3. Is the increase in FEV1 (and FVC) in children with asthma between 4-14 years of age with insufficient asthma control after inhalation of 400 μg SalbR different than after inhalation of 400 μg SalbG?
4. Is there a difference in the subjective feeling of the children after inhalation with 400 μg SalbR and after 400 μg SalbG, measured with a VAS score?

DETAILED DESCRIPTION:
Since 2016, pediatricians have regularly seen children with an asthma exacerbation, in which case salbutamol Sandoz was used as rescue medication in case of dyspnoea. The subjective impression is often that these children responded less well to this preparation in comparison to before or to the reference product, Ventolin.

After switching from the reference product (Ventolin, Salbutamol Reference, SalbR) to generic Salbutamol Sandoz (Salbutamol Generic, SalbG), parents also regularly spontaneously reported that they had the impression of reduced efficacy of SalbG.

Lareb received a striking number of reports in 2016 (63 of which 40 were reports concerning children) regarding an alleged reduced effect of SalbG compared to previous (reference) products containing salbutamol, such as Ventolin and Airomir. These reports mainly came after SalbG became the preferred drug of the Dutch health insurers.

In 2015, the concentration of SalbG in the aerosol dose doubled, whilst the release in micrograms would have remained the same, and oleic acid was added (as is also present in other dose aerosols).Reports received by Lareb came from both healthcare providers and (parents of) patients and did not clearly decrease in the course of 2016. An inventory via social media by the "LongFonds" clearly displayed the perception of lower efficacy amongst children as well as adults. This also led to a column in the broadcast of EenVandaag.

The CBG has studied and investigated the reports and signals, but has concluded that the quality control as carried out by the EMA was not a reason to remove Salbutamol Sandoz from the market. Various insurers have since accepted other generic products containing salbutamol in dose aerosol as an alternative instead of SalbG.

According to our information, there is currently no other party that will initiate a further in vivo efficacy study of SalbG. Pediatricians suspect Salbutamol Sandoz is less effective than the reference product, thus creating uncertainty and insufficiënt confidence regarding the quality of the product. However, this is essential as patients, parents and healthcare providers must be able to rely on the effectiveness of the "rescue medication".

The investigators consider it conceivable that a different composition of a dose aerosol can lead to a larger particle size (MMAD) and reduced lung deposition. Due to the lower suction power of children, this difference could especially occur with the first 100 microgram inhalation. In other words, the shape of the flow-volume curve differs between children. However, children may also react differently to the full 400 microgram dose.

The investigators also consider it conceivable that the registration requirements set by the EMA for the properties of a generic dose aerosol are not strict enough when it comes to administration to children, especially because the product has not been studied in the target group: children with acute asthma. For European registration of generic dose aerosols, it is sufficient if the MMAD particle size is within a range comparable to that of the reference product, and when the biological equivalence (plasma levels) is within a range equal to that of the reference product. The latter is often tested in a small group of healthy adult subjects. According to the EMA, the registration of a generic inhalation medication for children does not require that the efficacy in vivo (lung function, airway patency) or the bioavailability in children with (acute) asthma be investigated.

SalbG is the most commonly prescribed rescue drug in the Netherlands, so it is likely that many patients experiencing an asthma exacerbation use SalbG. It is therefore unclear whether SalbG is less effective than SalbR, or whether there must be another explanation for the reports.

The investigators consider it necessary for responsible care that rescue medication in children should be proven to be effective in the rescue setting. To gain clarity regarding the effectiveness of SalbG compared to SalbR, an in vivo study should be conducted in the target group, children with reduced asthma control.

The hypothesis of this study is that the reference product SalbR is more effective than SalbG in improving lung function in children with asthma, and that this difference is greater the more severe the airway resistance is. (Null hypothesis: there is no difference).

This could be explained by different properties and deposition of the aerosol.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent both parents in case of children aged < 12 years, informed consent both parents and patient of children aged 12-14 years
* Patients classified as doctor's diagnosed asthma, preferably with confirmed bronchial hyperreactivity or reversibility (FEV1 > 9% predicted) in earlier lung function assessment and/or known efficacy of salbutamol as rescue medication (either subjective or clinically)
* Indication for lung function assessment as part of regular medical care
* A score of < 20 on the C-ACT (children astma control questionnaire, 4-11 years) or ACT (12-16 years) and/or FEV1 <10% when compared to personal's best and/or FEV1 < 80% predicted and/or actual subjective impression of dyspnea in such severity that patient or caretaker would normally have used their bronchusdilatator

Exclusion Criteria:

* Status asthmaticus with a need for (continuous) nebulisation of salbutamol
* Inability of performing a technically adequate and reliable lung function assessment
* Inability of adequate instruction of patient and/or caretakers due to difficulty in communication and/or language barrier
* Clinically relevant comorbidities with impact on the lung function assessment (eg (cardio)pulmonary disease, muscle disease etc)

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
FEV1 (%) 100ug salbutamol | baseline
  FEV1 (%) after inhalation of 100 microgram salbutamol

SECONDARY OUTCOMES:
VAS 100ug salbutamol | baseline
  VAS score after inhalation of 100 microgram salbutamol
FEV1 (%) 400ug salbutamol | baseline
  FEV1 (%) after inhalation of 400 microgram salbutamol
VAS 400ug salbutamol | baseline
  VAS score after inhalation of 400 microgram salbutamol

OTHER OUTCOMES:
Age | baseline
  Age (years)
Length | baseline
  Length (cms)
Weight | baseline
  Weight (kgs)
Gender | baseline
  Gender (F/M)
Allergies | baseline
  Any known allergies
Inhalation corticosteroids (ICs) | baseline
  Use of inhalation corticosteroids (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No